CLINICAL TRIAL: NCT04496934
Title: Physical Activity as Adjunct Treatment for Opioid Substitution Therapy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); Kristiania University College (Other); University of Bergen (Other); Western Norway University of Applied Sciences (Other); Solli Distriktspsykiatriske Senter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/00731
Record Dates: First submitted 2018-10-25; First posted 2020-08-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder; Substance Use Disorders; Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Exercise intervention
  Interventions: Behavioral: Exercise
- Control (Active Comparator): The control group is a waiting list group. The participants will receive exercise intervention after twelve weeks of treatment as usual.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise of choice with a training contact: 3 hrs/week, total of 12 weeks.

SUMMARY:
In terms of research, it is documented that exercise has a positive effect on mental disorders. Studies have shown positive correlations between physical and mental health, also among substance users. Such a study has never been performed on patients in opioid substitution therapy (OST). Documentation on the physical health of patients and the effect of exercise is very limited. Treatment of substance users is a research area with insufficient knowledge about certain treatment effects. It is important that a treatment can both support and promote the user's own resources and efforts to change their habits of substance use.

The objective of this project is to examine the effect of exercise for OST patients, measured in relation to cognitive function and physical form. The target group consists of OST patients from 18 years of age and up, of both sexes, and on stable medication. At least 60 participants should complete the project, which is designed as a controlled randomized study (RCT). Participants in the intervention group start to exercise immediately after baseline testing. Participants in the control group are on a waiting list and will start to exercise after twelve weeks. Both groups undergo testing at baseline, after three, six and 12 months. Testing consists of two parts: A battery of cognitive and psychosocial assessments and an assessment of physical variables.

The research questions of this project are important in a public health perspective. Generated knowledge can be quickly applied to local treatment institutions in Norway.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign a informed consent form
* Must be participating in an opioid substitution program
* Must be on a steady fixed dose of medication
* Must be at least 18 years of age

Exclusion Criteria:

* Pregnancy
* Being in opioid substitution program for less than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Height and weight | 12 weeks
  Weight and height will be combined to report BMI in kg/m^2
Endurance | 12 weeks
  Ventilatory threshold/VO2max (endurance test on treadmill)
Strength | 12 weeks
  Push-ups (maximal test where the participants perform a maximum number of correct push-ups)
Balance | 12 weeks
  Stork Balance Test (timed test where the goal is to keep one's balance as long as possible)

SECONDARY OUTCOMES:
Alcohol use | 12 weeks
  AUDIT-E
Drug use | 12 weeks
  DUDIT-E
Executive functions | 12 weeks
  Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A)
Satisfaction with life | 12 weeks
  Satisfaction With Life Scale (SWLS)
  Values/scores:
  * 7 - Strongly agree
  * 6 - Agree
  * 5 - Slightly agree
  * 4 - Neither agree nor disagree
  * 3 - Slightly disagree
  * 2 - Disagree
  * 1 - Strongly disagree
  Results (sum of scores/values):
  31 - 35 Extremely satisfied 26 - 30 Satisfied 21 - 25 Slightly satisfied 20 Neutral 15 - 19 Slightly dissatisfied 10 - 14 Dissatisfied 5 - 9 Extremely dissatisfied The higher the score the better the outcome.
Sleep quality | 12 weeks
  Pittsburgh Sleep Quality Index (PSQI)
Attention | 12 weeks
  Connors Continuous Performance Test (CPT 3)

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir Mamen, PhD, Study Director — Kristiania University College; Lars Thore Fadnes, PhD, Study Director — University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT04496934/Prot_000.pdf
  • Informed Consent Form (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT04496934/ICF_001.pdf